CLINICAL TRIAL: NCT04890080
Title: Improvement of Resting Heart Rate After Exercise Training and Its Predictors in Chronic Obstructive Pulmonary Diseases
Brief Title: Resting Heart Rate in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ilknur Naz, Assoc. Prof., Izmir Katip Celebi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IKC111
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Pulmonary Rehabilitation; Exercise; COPD; Resting Heart Rate
Keywords: resting heart rate; COPD; exercise; pulmonary rehabilitation
MeSH Terms: conditions — Motor Activity; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PR Group (Experimental): Patients diagnosed with COPD according to GOLD and completed the 2-day / 8-week PR program
  Interventions: Other: Pulmonary Rehabilitation

INTERVENTIONS:
Other: Pulmonary Rehabilitation — Exercise training consisted of supervised breathing, aerobic, strengthening and stretching exercises for 8 weeks, 2 days a week. Breathing exercises included pursed lip, diaphragmatic, thoracic expansion and basal expansion exercises. Strength training included the lower and upper extremities, and it was performed 8-10 repetitions, either against gravity or using free weight, according to patient tolerance.

SUMMARY:
110 COPD patients who were participated in the PR program were included in the study. Resting Heart Rate , pulmonary functions, functional capacity, perception of dyspnea, quality of life and psychological symptoms compared before and after PR.

DETAILED DESCRIPTION:
In many studies, it has been reported that baroreceptor activity and heart rate variability decrease and resting heart rate (RHR) increases in COPD patients due to changes in cardiac autonomic function. Among the recommendations regarding pulmonary rehabilitation (PR) and exercise training in COPD patients, approaches such as including practices targeting RHR and developing implementation strategies that improve the cardiovascular system are recommended. The primary aim of our study is to examine the effect of comprehensive exercise training consisting of breathing, aerobic and strengthening exercises on RHR in COPD patients, and secondarily to determine the factors that affect RHR change after PR in COPD patients.

110 COPD patients who were participated in the PR program were included in our retrospective study. Resting Heart Rate , pulmonary functions, functional capacity, perception of dyspnea, quality of life and psychological symptoms compared before and after PR.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with COPD according to GOLD and completed the 2-day / 8-week PR program

Exclusion Criteria:

* With cardiovascular disease
* With additional diseases such as diabetes
* Receiving medical treatment that affects the autonomic nervous system
* Patients receiving long-term oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Resting Heart Rate | 1 minute
  number of beats per minute

SECONDARY OUTCOMES:
Functional Capacity | Change from baseline six minute walk distance at 8 week
  Six Minute- walk test
Dyspnea Assessment | Change from baseline dyspnea at 8 week
  Medical Research Council Scale(MRC); the MRC dyspnea scale is a questionnaire that consists of five statements about perceived breathlessness. (min 1- max 5 point) Higher scores mean a worse outcome.
Quality of Life Assessment | Change from baseline dyspnea at 8 week
  St. George Respiratory Questionnaire; Scores range from 0 to 100, with higher scores indicating more limitations.
Anxiety and Depression | Change from baseline dyspnea at 8 week
  Hospital Anxiety and Depression (HAD); The HADS questionnaire has seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.

IPD SHARING:
Plan to Share IPD: No